CLINICAL TRIAL: NCT05092581
Title: A Phase 1b, Open-Label, Single Dose Study Assessing the Pharmacokinetics, Safety, Tolerability, and Efficacy of Intravenous Anti-Spike(s) SARS-CoV-2 Monoclonal Antibodies (Casirivimab+Imdevimab) for the Treatment of Pediatric Patients Hospitalized Due to COVID-19
Brief Title: COVID-19 Study of Pharmacokinetics, Safety, Tolerability, and Efficacy of Intravenous Anti-Spike(s) SARS-CoV-2 Monoclonal Antibodies (Casirivimab+Imdevimab) for the Treatment of Pediatric Patients Hospitalized Due to COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Emerging SARS-CoV-2 variants impacting susceptibility to study drug
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R10933-10987-COV-2114; 2021-004535-84 (EudraCT Number)
Record Dates: First submitted 2021-10-22; First posted 2021-10-25 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: COVID-19
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-COV-2); coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — casirivimab and imdevimab drug combination; casirivimab; imdevimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- casirivimab+imdevimab (Experimental)
  Interventions: Drug: casirivimab+imdevimab

INTERVENTIONS:
Drug: casirivimab+imdevimab — Single dose weight-based equivalent administered intravenously (IV)
  Other Names: REGN-COV2; REGN10933; REGN10987; REGEN-COV™; Ronapreve™

SUMMARY:
The primary objectives of the study are:

* To characterize the concentrations of casirivimab+imdevimab in serum over time
* To evaluate the safety and tolerability of casirivimab+imdevimab

The secondary objective of the study is:

• To assess the immunogenicity of casirivimab+imdevimab

ELIGIBILITY:
Key Inclusion Criteria:

1. Has SARS-CoV-2 positive antigen or molecular diagnostic test ≤72 hours prior to study enrollment Note: historical record of positive result is acceptable as long as the sample was collected ≤72 hours prior to enrollment
2. Has symptoms consistent with COVID-19, as determined by the investigator, with onset ≤ 14 days before dosing
3. Hospitalized due to COVID-19
4. Provide informed consent signed by study patient or legally acceptable representative/guardian

Key Exclusion Criteria:

1. In the opinion of the investigator, unlikely to survive for >96 hours from screening
2. Neonates having gestational age of <29 weeks and weight <1.1 kg
3. Receiving extracorporeal membrane oxygenation (ECMO)
4. Has new-onset stroke or seizure disorder during hospitalization
5. Initiated on renal replacement therapy due to COVID-19
6. Has circulatory shock requiring vasopressors on dosing day Note: Patients who require vasopressors for sedation-related hypotension or reasons other than circulatory shock may be eligible in this study
7. Participation in a clinical research study, including any double-blind study, evaluating an investigational product within 30 days and less than 5 half-lives of the investigational product prior to the screening visit
8. Members of the clinical site study team and/or their immediate family
9. Plans to receive an investigational or approved SARS-CoV-2 vaccine within 90 days after study drug administration based on current Centers for Disease Control vaccination guidelines (CDC, 2021). Refer to the latest CDC guidance for any updates.

   Note: Patients who have already completed vaccination prior to study enrollment may be allowed in the study.
10. Prior use (within 90 days prior to study drug administration) or current use of any investigational, authorized, or approved passive antibody for prophylaxis of SARS-CoV-2 infection, including convalescent plasma, convalescent sera, hyperimmune globulin, or other monoclonal antibodies (eg, bamlanivimab and etesevimab, sotrovimab)

Note: Other protocol defined Inclusion/ Exclusion criteria apply

Ages: 1 Minute to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Concentrations of casirivimab+imdevimab in serum over time | Through day 169
Proportion of patients with treatment-emergent serious adverse events (SAEs) | Through day 29
Proportion of patients with infusion-related reactions | Through day 4
Proportion of patients with hypersensitivity reactions | Through day 29

SECONDARY OUTCOMES:
Incidence of anti-drug antibodies (ADA) to casirivimab+imdevimab over time | Through day 169
Incidence of neutralizing antibodies (NAb) to casirivimab+imdevimab over time | Through day 169

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - State University of New York at Stony Brook, Stony Brook, New York
  - Le Bonheur Children's Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/